CLINICAL TRIAL: NCT04317599
Title: A Retrospective Non Interventional Study on First Line Treatment for Patients With BRAFV600E Mutant Metastatic Colorectal Cancer (mCRC)
Acronym: CAPSTAN CRC
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Other Study IDs: NIS-PF0-2020-3141
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: BRAF V600E Mutation Positive; Metastatic Colorectal Cancer
Keywords: first line; retrospective study; mCRC; BRAF V600E
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non interventional: All BRAFV600E mutant patients having initiated a first-line treatment for mCRC between 01 January, 2016 and 31 December, 2018 (both days inclusive) with drugs registered for mCRC in respective country
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional — All BRAFV600E mutant patients having initiated a first-line treatment for mCRC between 01 January, 2016 and 31 December, 2018 (both days inclusive) with drugs registered for mCRC in respective country

SUMMARY:
The presence of a BRAFV600E mutation is considered a marker of poor prognosis in patients with mCRC, and findings from clinical trials have largely remained inconclusive regarding the efficacy of first line treatments for BRAF-mutant mCRC patients. In the absence of targeted/specific treatment for BRAF-mutant mCRC, treatment practices can vary based on local practices and guidelines. There is, therefore, an unmet need to document the current practices for first-line treatment of BRAF-mutant mCRC, and their effectiveness and safety in a real-world setting.

This real-world, multicenter non-interventional study (NIS) will describe the treatment patterns, effectiveness and safety of current treatment regimens in BRAFV600E mutant mCRC patients in Europe, with the aim to put the clinical study findings of the ongoing Phase 2, single-arm, open label trial (ANCHOR) into context of the current treatment landscape excluding investigational therapies. Additionally, the NIS output may be used to support future health technology assessment submissions and publications.

DETAILED DESCRIPTION:
This retrospective, multi-center longitudinal study on BRAFV600E mutant mCRC patients will be conducted in Europe to characterize the first-line treatment patterns. All BRAFV600E mutant patients having initiated a first-line treatment for mCRC between January 1st, 2016 and December 31st, 2018 (both days inclusive) with drugs registered for mCRC in respective country will be eligible to participate. The study will not provide or recommend any treatment or procedure; all decisions regarding treatment are made at the sole discretion of the treating physician in accordance with their usual practices and all eligible patients will be considered for enrollment.

The target countries for patient enrollment will include Germany, France, Italy, United Kingdom, Spain, Belgium, Austria and the Netherlands. Approximately 300 adult patients (≥18 years) from a mix of academic and non-academic sites (up to 65 sites) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed CRC that is metastatic and unresectable
* Presence of BRAFV600E mutation in tumor tissue, as confirmed by a local assay
* Initiated first-line treatment with drugs registered for mCRC in the respective country at the time of treatment between January 1st, 2016 and December 31st, 2018 (both days inclusive)
* Provision of informed consent or non-opposition to the patient (or next of kin, if applicable) for the use of data, according to local regulations

Exclusion Criteria:

Patients will be excluded from the study if they fulfil any of the following criteria:

* Patients with another concomitant cancer at the time of diagnosis*
* Patients participating in interventional trials on investigational drugs at the time of initiation of first-line treatment

  * Except for non-metastatic non-melanoma skin cancers, or in situ or benign neoplasms; a cancer will be considered concomitant if it occurs within 5 years of mCRC diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with BRAFV600E mutant mCRC (determined by local laboratory result) in the target countries and initiating first line treatment between January 1st, 2016 and December 31st, 2018 (both days inclusive) will be eligible for enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Asselain, MD, PhD, Study Chair; Dirk Arnold, MD, PhD, Study Chair; Erika Martinelli, MD, PhD, Study Chair
Locations (34):
- Austria (2):
  - Barmherzige Brüder Krankenhaus St. Veit/Glan., Saint Veit/Glan
  - Medizinische Universität Wien, Vienna
- Belgium (4):
  - Imelda VZW, Bonheiden
  - AZ Klina, Brasschaat
  - UZ Leuven, Leuven
  - CHC MontLégia, Liège
- France (8):
  - CHRU de Besançon, Besançon
  - GHPSO (Groupe Hospitalier Sud de l'Oise), Creil
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Franco-Britannique, Levallois-Perret
  - Centre Oscar Lambert, Lille
  - ICM Val d'Aurelle, Montpellier
  - CHU de Poitiers, Poitiers
  - Gustave Roussy, Villejuif
- Germany (7):
  - Klinikum Aschaffenburg Medical Klinik IV, Aschaffenburg
  - Studienzentrale Gokos, Dresden
  - Universitätsklinikum Essen, Essen
  - Facharztzentrum Eppendorf, Hamburg
  - Oncoresearch Lerchenfeld, Hamburg
  - MVZ Mitte Leipzig, Leipzig
  - MZ Onkologie Velbert/Ratingen/Mettmann, Velbert
- Italy (6):
  - Clinica Oncologica Ospedali Riuniti di Ancona, Ancona
  - Santa Maria Goretti Hospital, Latina
  - Instituto Nazionale Tumori, IRCCS, Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - AUSL-IRCCS of Reggio Emilia-Clinical Cancer Center, Reggio Emilia
  - Asst Valle Olona, Saronno
- Spain (3):
  - Hospital del Mar, Barcelona
  - La Paz University Hospital, Madrid
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Harrogate & District NHS Foundation Trust, Harrogate
  - Imperial College Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Interventional: All BRAFV600E mutant patients having initiated a first-line treatment for mCRC between 01 January, 2016 and 31 December, 2018 (both days inclusive) with drugs registered for mCRC in respective country
  Non Interventional study: Non Interventional study
Period: Overall Study
Arm/Group | Non Interventional
Started | 274
Completed | 255
Not Completed | 19
Not completed — ineligible due to inclusion/exclusion criteria | 15
Not completed — treatment outside standard of care | 4

BASELINE CHARACTERISTICS:
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Age, Customized [Count of Participants; unit: Participants]
  ≤ 60 years | 87
  61-70 years | 68
  > 70 years | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 106
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4
  Belgium | 28
  Italy | 52
  United Kingdom | 17
  France | 74
  Germany | 45
  Spain | 35
Anthropometry - Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.42 (5.44)
Disease stage at initial diagnosis [Count of Participants; unit: Participants] — TNM stage at initial diagnosis of colorectal cancer. Stage I: Cancer is still in the inner lining, but has grown through the mucosa of the colon and invaded the muscle layer.
  Stage II: The cancer has grown beyond the mucosa of the colon but has not spread to the lymph nodes Stage III: The cancer has spread to the lymph nodes near the colon, it has not spread further.
  Stage IV: The cancer has spread outside of the colon and has been carried through the lymph and blood systems to distant parts of the body, this is known as metastasis. Population: Data not available for all patients.
  Participants
    number analyzed (Participants) | 226
    I | 4
    II | 24
    III | 48
    IV | 150
Histology at initial diagnosis [Count of Participants; unit: Participants] — Population: Data not available for all patients.
  Participants
    number analyzed (Participants) | 253
    Adenocarcinoma | 252
    Other carcinoma | 1
Primary tumor location [Count of Participants; unit: Participants]
  left and/or rectum | 83
  right only | 134
  other (left and right or transverse or right and rectum or not applicable) | 38
Number of metastatic sites [Count of Participants; unit: Participants]
  1 site | 115
  2 sites | 82
  ≥3 sites | 58
Characterization of metastasis [Mean (Standard Deviation); unit: months] — Diagnosis of metastatic CRC after CRC diagnosis
  months | 4.75 (12.25)
Location of metastasis [Count of Participants; unit: Participants]
  Liver | 148
  Liver only | 48
  Lungs | 68
  Lymph nodes | 89
  Bone | 8
  Peritoneum | 112
  Central Nervous System | 2
  Abdomen (including 7 patients with "ovaries") | 12
  Other | 25
Performance Status [Count of Participants; unit: Participants] — ECOG: Eastern Cooperative Oncology Group ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG = 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Population: ECOG performance status score at mCRC diagnosis was recorded for 150 patients
  Participants
    number analyzed (Participants) | 150
    ECOG 0 | 80
    ECOG 1 | 56
    ECOG 2 | 10
    ECOG 3 | 4
Patients with at least one comorbidity [Count of Participants; unit: Participants] — Population: Data not available for all patients.
  Participants
    number analyzed (Participants) | 253
    (all) | 129
Number of comorbidities [Mean (Standard Deviation); unit: comorbidities] — Population: Data not available for all patients.
  comorbidities
    number analyzed (Participants) | 253
    (all) | 0.8 (1.0)
Types of comorbidity [Count of Participants; unit: Participants] — Population: Data not available for all patients.
  Participants
    Treated hypertension: number analyzed (Participants) | 253
    Treated hypertension | 100
    Heart rhythm disorder: number analyzed (Participants) | 253
    Heart rhythm disorder | 19
    Peripheral vascular disease: number analyzed (Participants) | 253
    Peripheral vascular disease | 15
    Ischemic cardiac disorder: number analyzed (Participants) | 253
    Ischemic cardiac disorder | 12
    Chronic pulmonary disease: number analyzed (Participants) | 253
    Chronic pulmonary disease | 12
    Rheumatic or connective tissue disease: number analyzed (Participants) | 253
    Rheumatic or connective tissue disease | 12
    Diabetes mellitus with end-organ damage: number analyzed (Participants) | 253
    Diabetes mellitus with end-organ damage | 9
    Moderate or severe liver disease: number analyzed (Participants) | 253
    Moderate or severe liver disease | 6
    Congestive heart failure: number analyzed (Participants) | 253
    Congestive heart failure | 4
    Moderate or severe renal disease: number analyzed (Participants) | 253
    Moderate or severe renal disease | 4
    Cerebrovascular disease: number analyzed (Participants) | 253
    Cerebrovascular disease | 1
    Acquired immunodeficiency syndrome (AIDS): number analyzed (Participants) | 253
    Acquired immunodeficiency syndrome (AIDS) | 1
1st line therapy received for the mCRC [Count of Participants; unit: Participants]
  monotherapy +/- Targeted Therapy (TT) | 17
  Doublet chemotherapy (CT) | 72
  Doublet CT + TT | 118
  Triplet CT | 8
  Triplet CT + TT | 40
Number of patients with at least one surgery for either CRC or mCRC [Count of Participants; unit: Participants] | 163
Number of patients receiving radiotherapy for CRC or mCRC [Count of Participants; unit: Participants] | 29
Number of patients with at least one SACT (Systemic anti-cancer therapy) treatment [Count of Participants; unit: Participants] — Population: Analysis done for 254 patients
  Participants
    number analyzed (Participants) | 254
    (all) | 40
RAS testing [Count of Participants; unit: Participants] — Test of changes (mutations) in a group of genes called RAS genes Population: 234 patients had at least one RAS testing.
  Participants
    number analyzed (Participants) | 234
    Mutated | 16
    Wild type | 217
    Unknown | 1
Method of RAS testing [Count of Participants; unit: Participants] — Population: 230 patients had this information available.
  Participants
    number analyzed (Participants) | 230
    Next generation sequencing (NGS) | 89
    Polymerase chain reaction (PCR) | 81
    Other | 60
Microsatellite instability (MSI) testing [Count of Participants; unit: Participants] — Microsatellite instability refers to a change that occurs in certain cells (such as cancer cells) in which the number of repeated DNA bases in a microsatellite (a short, repeated sequence of DNA) is different from what it was when the microsatellite was inherited.
  MSI testing is used to classify CRC tumors as MSI-high (MSI-H), MSI-low, and microsatellite stable tumors. Population: 153 patients had at least one MSI testing.
  Participants
    number analyzed (Participants) | 153
    MSI low | 10
    MSI stable | 103
    MSI high | 36
    MSI unknown | 4
MMR gene (if MSI was measured) [Count of Participants; unit: Participants] — Testing to check for changes in any of the mismatch repair (MMR) genes (MLH1, MSH2, MSH6, and PMS2). Population: 119 patients had this information available.
  Participants
    number analyzed (Participants) | 119
    dMMR | 29
    pMMR | 90
Serum albumin levels [Mean (Standard Deviation); unit: g/dL] — Population: Data not available for all patients.
  g/dL
    number analyzed (Participants) | 96
    (all) | 10.17 (14.43)
Hemoglobin levels [Mean (Standard Deviation); unit: g/dL] — Population: Data not available for all patients.
  g/dL
    number analyzed (Participants) | 167
    (all) | 11.93 (1.91)
Hemoglobin levels - normal/abnormal [Count of Participants; unit: Participants] — Population: Data not available for all patients.
  Participants
    number analyzed (Participants) | 167
    Abnormal | 79
    Normal (between [12 ;16] g/dL) | 88
Platelet levels [Mean (Standard Deviation); unit: 10^9 platelets/L] — Population: Data not available for all patients.
  10^9 platelets/L
    number analyzed (Participants) | 166
    (all) | 342.64 (142.86)
Leucocyte levels [Mean (Standard Deviation); unit: 10^9 cells/L] — Population: Data not available for all patients.
  10^9 cells/L
    number analyzed (Participants) | 165
    (all) | 9.07 (3.33)
Neutrophil (absolute count) [Mean (Standard Deviation); unit: 10^9 cells/L] — Population: Data not available for all patients.
  10^9 cells/L
    number analyzed (Participants) | 151
    (all) | 6.19 (2.96)
Neutrophil (differential count) [Mean (Standard Deviation); unit: percentage of total blood cells] — Population: Data not available for all patients.
  percentage of total blood cells
    number analyzed (Participants) | 145
    (all) | 67.75 (11.77)
C-reactive protein levels [Mean (Standard Deviation); unit: mg/L] — Population: This data was not available for all patients.
  mg/L
    number analyzed (Participants) | 61
    (all) | 13.99 (12.45)
Carcinoembryonic antigen (CEA) levels [Mean (Standard Deviation); unit: ng/mL] — Population: This data was not available for all patients.
  ng/mL
    number analyzed (Participants) | 109
    (all) | 16.20 (18.46)
Carbohydrate antigen 19-9 (CA 19.9) levels [Mean (Standard Deviation); unit: U/mL] — Population: This data was not available for all patients.
  U/mL
    number analyzed (Participants) | 79
    (all) | 149.18 (220.75)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Patterns for First-line Systemic Anticancer Therapy (SACT) in BRAFV600E Mutant mCRC Patients
Description: First-line SACT treatment patterns in BRAFV600E mutant mCRC patients described by agent or combination of agents received
Time Frame: time from treatment initiation (for mCRC) up to 31 December 2020
Population: *treated as doublet CT + anti-EGFR for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Participants
  Monotherapy +/- targetted therapy (TT) | 17
  Monotherapy +/- TT : : Fluropyrimidine monotherapy | 6
  Monotherapy +/- TT : : Fluropyrimidine monotherapy / Bevacizumab | 10
  Monotherapy +/- TT : : Fluropyrimidine monotherapy / Panitumumab | 1
  Doublet chemotherapy (CT) | 72
  Doublet CT : : CAPOX | 11
  Doublet CT : : FOLFIRI | 7
  Doublet CT : : FOLFOX | 49
  Doublet CT : : Fluoropyrimidine + (Irinotecan or Folic Acid) | 3
  Doublet CT : : XELIRI | 2
  Doublet CT + TT | 118
  Doublet CT + TT : Doublet CT + anti-VEGF | 99
  Doublet CT + TT : Doublet CT + anti-VEGF : CAPOX / Bevacizumab | 8
  Doublet CT + TT : Doublet CT + anti-VEGF : FOLFIRI / Aflibercept | 2
  Doublet CT + TT : Doublet CT + anti-VEGF : FOLFIRI / Bevacizumab | 20
  Doublet CT + TT : Doublet CT + anti-VEGF : FOLFOX / Bevacizumab | 69
  Doublet CT + TT : Doublet CT + anti-EGFR | 19
  Doublet CT + TT : Doublet CT + anti-EGFR : FOLFIRI / Cetuximab | 3
  Doublet CT + TT : Doublet CT + anti-EGFR : FOLFIRI / Panitumumab | 2
  Doublet CT + TT : Doublet CT + anti-EGFR : Tomiri / Panitumumab | 1
  Doublet CT + TT : Doublet CT + anti-EGFR : FOLFOX / Cetuximab | 5
  Doublet CT + TT : Doublet CT + anti-EGFR : FOLFOX / Panitumumab | 7
  Doublet CT + TT : Doublet CT + anti-EGFR : FOLFOX / Cetuximab + Avelumab* | 1
  Triplet CT | 8
  Triplet CT : : FOLFIRINOX | 2
  Triplet CT : : FOLFOXIRI | 6
  Triplet CT + TT | 40
  Triplet CT + TT : Triplet + anti-VEGF | 38
  Triplet CT + TT : Triplet + anti-VEGF : FOLFIRINOX / Bevacizumab | 4
  Triplet CT + TT : Triplet + anti-VEGF : FOLFOXIRI / Bevacizumab | 34
  Triplet CT + TT : Triplet + anti-EGFR | 2
  Triplet CT + TT : Triplet + anti-EGFR : FOLFOXIRI / Cetuximab | 1
  Triplet CT + TT : Triplet + anti-EGFR : FOLFOXIRI / Panitumumab | 1

2. Primary Outcome: Duration of Treatment for First-line Systemic Anticancer Therapy (SACT) in BRAFV600E Mutant mCRC Patients
Description: First-line SACT treatment patterns in BRAFV600E mutant mCRC patients described by Duration of Treatment
Time Frame: time from treatment initiation (for mCRC) up to 31 December 2020
Population: A total of 255 patients were included in the full analysis set (FAS). Data for 2 patients were not available.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Non Interventional
Number analyzed (Participants) | 253
months | 6.04 (5.79)

3. Primary Outcome: Switch in mCRC First-line Systemic Anticancer Therapy (SACT) Treatment in BRAFV600E Mutant mCRC Patients
Description: Switch in mCRC first-line SACT treatment in BRAFV600E mutant mCRC patients.
Time Frame: time from treatment initiation (for mCRC) up to 31 December 2020
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Participants
  Switch to other treatment | 80
  Switch to other treatment: maintenance | 30
  Reason for switch: toxicity | 24
  Reason for switch: lack of response | 13
  Reason for switch: other | 13
  Switch to: FOLFOX | 21
  Switch to: CAPOX | 1
  Switch to: FOLFIRI | 16
  Switch to: Fluoropyrimidine monotherapy | 27
  Switch to: FOLFOXIRI | 4
  Switch to: FOLFIRINOX | 3
  Switch to: Tomiri | 1
  Switch to: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 2
  Switch to: Other | 4
  Switch to: BRAFi + Other | 1
  If switch with FOLFOX, CAPOX, FOLFIRI, Fluoropyrimidine or FOLFIXIRI - | 53
  - then, in combination with: Panitumumab | 4
  - then, in combination with: Cetuximab | 1
  - then, in combination with: Bevacizumab | 48
  Switch regiment: BRAFi + Other | 1
  Switch regiment: CAPOX / Bevacizumab | 1
  Switch regiment: FOLFIRI | 6
  Switch regiment: FOLFIRI / Bevacizumab | 8
  Switch regiment: FOLFIRI / Cetuximab | 1
  Switch regiment: FOLFIRI / Panitumumab | 1
  Switch regiment: FOLFIRINOX | 2
  Switch regiment: FOLFIRINOX / Bevacizumab | 1
  Switch regiment: FOLFOX | 6
  Switch regiment: FOLFOX / Bevacizumab | 14
  Switch regiment: FOLFOX / Panitumumab | 1
  Switch regiment: FOLFOXIRI / Bevacizumab | 4
  Switch regiment: Fluoropyrimidine monotherapy | 6
  Switch regiment: Fluoropyrimidine monotherapy / Bevacizumab | 19
  Switch regiment: Fluoropyrimidine monotherapy / Panitumumab | 2
  Switch regiment: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 1
  Switch regiment: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 1
  Switch regiment: Other | 4
  Switch regiment: Tomiri | 1

4. Secondary Outcome: Demographic and Clinical Characteristics
Description: Description of the demographic and clinical profile of patients at the time of treatment initiation (for mCRC) TNM stage of colorectal cancer. Stage I: Cancer is still in the inner lining, but has grown through the mucosa of the colon and invaded the muscle layer.
  Stage II: The cancer has grown beyond the mucosa of the colon but has not spread to the lymph nodes Stage III: The cancer has spread to the lymph nodes near the colon, it has not spread further.
  Stage IV: The cancer has spread outside of the colon and has been carried through the lymph and blood systems to distant parts of the body, this is known as metastasis.
Time Frame: from the date of the start of first-line treatment for mCRC up to 31 December 2020
Population: Disease stage at initial diagnosis of CRC by first line treatment regimen Data were available for 226 of the 255 patients included in the FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 226
Participants
  Monotherapy +/- TT: number analyzed (Participants) | 15
  Monotherapy +/- TT: TNM Stage I | 0
  Monotherapy +/- TT: TNM Stage II | 3
  Monotherapy +/- TT: TNM Stage III | 4
  Monotherapy +/- TT: TNM Stage IV | 8
  Doublet CT: number analyzed (Participants) | 59
  Doublet CT: TNM Stage I | 1
  Doublet CT: TNM Stage II | 7
  Doublet CT: TNM Stage III | 10
  Doublet CT: TNM Stage IV | 41
  Doublet CT + TT: number analyzed (Participants) | 113
  Doublet CT + TT: TNM Stage I | 2
  Doublet CT + TT: TNM Stage II | 10
  Doublet CT + TT: TNM Stage III | 26
  Doublet CT + TT: TNM Stage IV | 75
  Triplet CT: number analyzed (Participants) | 6
  Triplet CT: TNM Stage I | 0
  Triplet CT: TNM Stage II | 0
  Triplet CT: TNM Stage III | 2
  Triplet CT: TNM Stage IV | 4
  Triplet CT + TT: number analyzed (Participants) | 33
  Triplet CT + TT: TNM Stage I | 1
  Triplet CT + TT: TNM Stage II | 4
  Triplet CT + TT: TNM Stage III | 6
  Triplet CT + TT: TNM Stage IV | 22

5. Secondary Outcome: Progression-free Survival (PFS)
Description: the length of time between initiation of first-line treatment for mCRC and the first documented disease progression or death.
  Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from the date of the start of first-line treatment for mCRC up to 31 December 2020
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
months | 5.98 [5.32 to 6.67]

6. Secondary Outcome: Overall Survival (OS)
Description: length of time between first-line treatment initiation (for mCRC) and death (due to any cause)
Time Frame: from the date of the start of first-line treatment for mCRC up to 31 December 2020
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
months | 12.68 [11.60 to 14.13]

7. Secondary Outcome: Overall Response Rate (ORR)
Description: complete response (CR) or partial response (PR), during the first line treatment Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: from the date of the start of first-line treatment for mCRC until the end of first-line treatment up to 31 December 2020
Population: Data were available for 221 of the 255 patients included in the FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 221
percentage of participants | 37.1 [30.7 to 43.5]

8. Secondary Outcome: Time to Treatment Cessation
Description: the length of time between initiation of first-line treatment for mCRC and documented disease progression (or start of subsequent Line Of Treatment (LOT), if disease progression is not well documented in patient medical record), treatment discontinuation or switch to another treatment (defined as change from one treatment regimen to another treatment regimen, e.g., change from FOLFOX-based regimen to FOLFIRI or irinotecan-based regimen)
Time Frame: from the date of the start of first-line treatment for mCRC until the documented disease progression up to 31 December 2020
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
months | 4.83 [4.01 to 5.32]

9. Secondary Outcome: Description of BRAF Mutation Testing Procedure in Regards With the First-line Treatment in BRAFV600E Mutant mCRC Patients
Description: Description of testing procedures of BRAF mutation testing since mCRC diagnosis and since first-line treatment for mCRC
Time Frame: as for outcome 7
Population: Data not available for all patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Participants
  Number of BRAF testing: 1 | 244
  Number of BRAF testing: 2 | 11
  Timing of 1st BRAF testing: before 1L (2 to 38 months before 1st line initiation): number analyzed (Participants) | 225
  Timing of 1st BRAF testing: before 1L (2 to 38 months before 1st line initiation) | 62
  Timing of 1st BRAF testing: before 1L (less than 2 months before 1st line initiation): number analyzed (Participants) | 225
  Timing of 1st BRAF testing: before 1L (less than 2 months before 1st line initiation) | 140
  Timing of 1st BRAF testing: during 1L: number analyzed (Participants) | 225
  Timing of 1st BRAF testing: during 1L | 21
  Timing of 1st BRAF testing: after 1L and before 2L: number analyzed (Participants) | 225
  Timing of 1st BRAF testing: after 1L and before 2L | 1
  Timing of 1st BRAF testing: during 2L: number analyzed (Participants) | 225
  Timing of 1st BRAF testing: during 2L | 1
  BRAF test sample: tumor sample | 252
  BRAF test sample: ctDNA | 3
  If tumor sample, tumor sample tested: archival: number analyzed (Participants) | 228
  If tumor sample, tumor sample tested: archival | 175
  If tumor sample, tumor sample tested: fresh: number analyzed (Participants) | 228
  If tumor sample, tumor sample tested: fresh | 53
  Method used: PCR: number analyzed (Participants) | 226
  Method used: PCR | 104
  Method used: NGS: number analyzed (Participants) | 226
  Method used: NGS | 86
  Method used: Other: number analyzed (Participants) | 226
  Method used: Other | 10
  Method used: high resolution melting: number analyzed (Participants) | 226
  Method used: high resolution melting | 4
  Method used: mass spectrometry: number analyzed (Participants) | 226
  Method used: mass spectrometry | 22

10. Secondary Outcome: Description of BRAF Mutation Testing Timing in Regards With the First-line Treatment in BRAFV600E Mutant mCRC Patients
Description: Time to BRAF mutation testing since mCRC diagnosis and since first-line treatment for mCRC
Time Frame: as for outcome 7
Population: Data not available for all patients.
Measure: Mean (Standard Error); unit: months
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
months
  Time from metastatic diagnosis to 1st BRAF mutation testing (if after metastatic diagnosis): number analyzed (Participants) | 157
  Time from metastatic diagnosis to 1st BRAF mutation testing (if after metastatic diagnosis) | 0.6 (1.7)
  Time from metastatic diagnosis to 1st BRAF mutation testing (if before metastatic diagnosis): number analyzed (Participants) | 66
  Time from metastatic diagnosis to 1st BRAF mutation testing (if before metastatic diagnosis) | 6.1 (7.9)

11. Other Pre Specified Outcome: Reasons for Alteration or Discontinuation of First-line Treatment in BRAFV600E Mutant mCRC Patients
Description: Description of reasons for alteration or discontinuation of first-line treatment for mCRC in BRAFV600E Mutant mCRC Patients
Time Frame: as for outcome 7
Population: *due to other reasons than progression or toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Participants
  Patient with treatment alteration: number analyzed (Participants) | 237
  Patient with treatment alteration | 137
  Most important reason for treatment alteration: Planned alteration: number analyzed (Participants) | 132
  Most important reason for treatment alteration: Planned alteration | 10
  Most important reason for treatment alteration: Toxicity: number analyzed (Participants) | 132
  Most important reason for treatment alteration: Toxicity | 100
  Most important reason for treatment alteration: Poor performance status of patient: number analyzed (Participants) | 132
  Most important reason for treatment alteration: Poor performance status of patient | 6
  Most important reason for treatment alteration: Other: number analyzed (Participants) | 132
  Most important reason for treatment alteration: Other | 16
  Patient with treatment discontinuation: number analyzed (Participants) | 251
  Patient with treatment discontinuation | 248
  Most important reason for treatment discontinuation: Progression: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Progression | 158
  Most important reason for treatment discontinuation: Toxicity: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Toxicity | 19
  Most important reason for treatment discontinuation: BRAF test available: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: BRAF test available | 5
  Most important reason for treatment discontinuation: Planned discontinuation: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Planned discontinuation | 21
  Most important reason for treatment discontinuation: Patient choice: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Patient choice | 6
  Most important reason for treatment discontinuation: Poor performance status of patient: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Poor performance status of patient | 16
  Most important reason for treatment discontinuation: Death*: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Death* | 4
  Most important reason for treatment discontinuation: Other: number analyzed (Participants) | 238
  Most important reason for treatment discontinuation: Other | 9

12. Other Pre Specified Outcome: Other Types of SACT Treatment Line Regiments After First-line Treatment for mCRC in BRAFV600E Mutant mCRC Patients
Description: Description of the types of treatments after first-line SACT treatment (2nd-line to 7th-line) in BRAFV600E Mutant mCRC Patients.
Time Frame: as for outcome 7
Population: Not all patients went through all lines of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Non Interventional
Number analyzed (Participants) | 255
Participants
  2nd: number analyzed (Participants) | 134
  2nd: BRAFi / Cetuximab | 7
  2nd: BRAFi / Cetuximab + Irinotecan | 4
  2nd: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 1
  2nd: BRAFi / MEKi / Cetuximab | 16
  2nd: BRAFi / MEKi / Panitumumab | 1
  2nd: CAPOX | 2
  2nd: Cetuximab monotherapy | 1
  2nd: FOLFIRI | 19
  2nd: FOLFIRI / Aflibercept | 7
  2nd: FOLFIRI / Bevacizumab | 20
  2nd: FOLFIRI / Cetuximab | 8
  2nd: FOLFIRI / Panitumumab | 5
  2nd: FOLFOX | 4
  2nd: FOLFOX / Bevacizumab | 7
  2nd: FOLFOX / Cetuximab | 1
  2nd: FOLFOX / Panitumumab | 3
  2nd: FOLFOXIRI | 1
  2nd: FOLFOXIRI / Bevacizumab | 6
  2nd: Fluoropyrimidine monotherapy | 1
  2nd: Fluoropyrimidine monotherapy / Bevacizumab | 2
  2nd: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 1
  2nd: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 1
  2nd: Irinotecan | 1
  2nd: Irinotecan / Cetuximab | 4
  2nd: Irinotecan / Panitumumab | 1
  2nd: Other | 7
  2nd: Panitumumab monotherapy | 2
  2nd: XELIRI / Bevacizumab | 1
  2nd: BRAFi | 0
  2nd: CAPOX / Bevacizumab | 0
  2nd: Fluoropyrimidine monotherapy / Panitumumab | 0
  2nd: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 0
  3rd: number analyzed (Participants) | 77
  3rd: BRAFi / Cetuximab | 2
  3rd: BRAFi / Cetuximab + Irinotecan | 5
  3rd: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  3rd: BRAFi / MEKi / Cetuximab | 6
  3rd: BRAFi / MEKi / Panitumumab | 2
  3rd: CAPOX | 0
  3rd: Cetuximab monotherapy | 1
  3rd: FOLFIRI | 2
  3rd: FOLFIRI / Aflibercept | 4
  3rd: FOLFIRI / Bevacizumab | 9
  3rd: FOLFIRI / Cetuximab | 2
  3rd: FOLFIRI / Panitumumab | 0
  3rd: FOLFOX | 4
  3rd: FOLFOX / Bevacizumab | 5
  3rd: FOLFOX / Cetuximab | 0
  3rd: FOLFOX / Panitumumab | 0
  3rd: FOLFOXIRI | 2
  3rd: FOLFOXIRI / Bevacizumab | 1
  3rd: Fluoropyrimidine monotherapy | 0
  3rd: Fluoropyrimidine monotherapy / Bevacizumab | 3
  3rd: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 0
  3rd: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  3rd: Irinotecan | 1
  3rd: Irinotecan / Cetuximab | 2
  3rd: Irinotecan / Panitumumab | 2
  3rd: Other | 20
  3rd: Panitumumab monotherapy | 1
  3rd: XELIRI / Bevacizumab | 0
  3rd: BRAFi | 1
  3rd: CAPOX / Bevacizumab | 1
  3rd: Fluoropyrimidine monotherapy / Panitumumab | 1
  3rd: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 0
  4th line: number analyzed (Participants) | 39
  4th line: BRAFi / Cetuximab | 0
  4th line: BRAFi / Cetuximab + Irinotecan | 2
  4th line: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  4th line: BRAFi / MEKi / Cetuximab | 3
  4th line: BRAFi / MEKi / Panitumumab | 0
  4th line: CAPOX | 0
  4th line: Cetuximab monotherapy | 1
  4th line: FOLFIRI | 1
  4th line: FOLFIRI / Aflibercept | 4
  4th line: FOLFIRI / Bevacizumab | 0
  4th line: FOLFIRI / Cetuximab | 1
  4th line: FOLFIRI / Panitumumab | 0
  4th line: FOLFOX | 4
  4th line: FOLFOX / Bevacizumab | 1
  4th line: FOLFOX / Cetuximab | 0
  4th line: FOLFOX / Panitumumab | 1
  4th line: FOLFOXIRI | 1
  4th line: FOLFOXIRI / Bevacizumab | 1
  4th line: Fluoropyrimidine monotherapy | 0
  4th line: Fluoropyrimidine monotherapy / Bevacizumab | 0
  4th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 0
  4th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  4th line: Irinotecan | 0
  4th line: Irinotecan / Cetuximab | 2
  4th line: Irinotecan / Panitumumab | 0
  4th line: Other | 15
  4th line: Panitumumab monotherapy | 1
  4th line: XELIRI / Bevacizumab | 0
  4th line: BRAFi | 0
  4th line: CAPOX / Bevacizumab | 0
  4th line: Fluoropyrimidine monotherapy / Panitumumab | 1
  4th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 0
  5th line: number analyzed (Participants) | 14
  5th line: BRAFi / Cetuximab | 0
  5th line: BRAFi / Cetuximab + Irinotecan | 2
  5th line: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  5th line: BRAFi / MEKi / Cetuximab | 1
  5th line: BRAFi / MEKi / Panitumumab | 0
  5th line: CAPOX | 0
  5th line: Cetuximab monotherapy | 0
  5th line: FOLFIRI | 0
  5th line: FOLFIRI / Aflibercept | 1
  5th line: FOLFIRI / Bevacizumab | 0
  5th line: FOLFIRI / Cetuximab | 0
  5th line: FOLFIRI / Panitumumab | 0
  5th line: FOLFOX | 0
  5th line: FOLFOX / Bevacizumab | 0
  5th line: FOLFOX / Cetuximab | 0
  5th line: FOLFOX / Panitumumab | 0
  5th line: FOLFOXIRI | 0
  5th line: FOLFOXIRI / Bevacizumab | 0
  5th line: Fluoropyrimidine monotherapy | 0
  5th line: Fluoropyrimidine monotherapy / Bevacizumab | 0
  5th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 0
  5th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  5th line: Irinotecan | 0
  5th line: Irinotecan / Cetuximab | 0
  5th line: Irinotecan / Panitumumab | 0
  5th line: Other | 8
  5th line: Panitumumab monotherapy | 1
  5th line: XELIRI / Bevacizumab | 0
  5th line: BRAFi | 0
  5th line: CAPOX / Bevacizumab | 0
  5th line: Fluoropyrimidine monotherapy / Panitumumab | 0
  5th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 1
  6th line: number analyzed (Participants) | 5
  6th line: BRAFi / Cetuximab | 0
  6th line: BRAFi / Cetuximab + Irinotecan | 0
  6th line: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  6th line: BRAFi / MEKi / Cetuximab | 0
  6th line: BRAFi / MEKi / Panitumumab | 0
  6th line: CAPOX | 0
  6th line: Cetuximab monotherapy | 1
  6th line: FOLFIRI | 0
  6th line: FOLFIRI / Aflibercept | 0
  6th line: FOLFIRI / Bevacizumab | 0
  6th line: FOLFIRI / Cetuximab | 0
  6th line: FOLFIRI / Panitumumab | 0
  6th line: FOLFOX | 2
  6th line: FOLFOX / Bevacizumab | 0
  6th line: FOLFOX / Cetuximab | 0
  6th line: FOLFOX / Panitumumab | 0
  6th line: FOLFOXIRI | 0
  6th line: FOLFOXIRI / Bevacizumab | 0
  6th line: Fluoropyrimidine monotherapy | 1
  6th line: Fluoropyrimidine monotherapy / Bevacizumab | 0
  6th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 0
  6th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  6th line: Irinotecan | 0
  6th line: Irinotecan / Cetuximab | 0
  6th line: Irinotecan / Panitumumab | 1
  6th line: Other | 0
  6th line: Panitumumab monotherapy | 0
  6th line: XELIRI / Bevacizumab | 0
  6th line: BRAFi | 0
  6th line: CAPOX / Bevacizumab | 0
  6th line: Fluoropyrimidine monotherapy / Panitumumab | 0
  6th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 0
  7th line: number analyzed (Participants) | 1
  7th line: BRAFi / Cetuximab | 1
  7th line: BRAFi / Cetuximab + Irinotecan | 0
  7th line: BRAFi+ Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  7th line: BRAFi / MEKi / Cetuximab | 0
  7th line: BRAFi / MEKi / Panitumumab | 0
  7th line: CAPOX | 0
  7th line: Cetuximab monotherapy | 0
  7th line: FOLFIRI | 0
  7th line: FOLFIRI / Aflibercept | 0
  7th line: FOLFIRI / Bevacizumab | 0
  7th line: FOLFIRI / Cetuximab | 0
  7th line: FOLFIRI / Panitumumab | 0
  7th line: FOLFOX | 0
  7th line: FOLFOX / Bevacizumab | 0
  7th line: FOLFOX / Cetuximab | 0
  7th line: FOLFOX / Panitumumab | 0
  7th line: FOLFOXIRI | 0
  7th line: FOLFOXIRI / Bevacizumab | 0
  7th line: Fluoropyrimidine monotherapy | 0
  7th line: Fluoropyrimidine monotherapy / Bevacizumab | 0
  7th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) | 0
  7th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Cetuximab | 0
  7th line: Irinotecan | 0
  7th line: Irinotecan / Cetuximab | 0
  7th line: Irinotecan / Panitumumab | 0
  7th line: Other | 0
  7th line: Panitumumab monotherapy | 0
  7th line: XELIRI / Bevacizumab | 0
  7th line: BRAFi | 0
  7th line: CAPOX / Bevacizumab | 0
  7th line: Fluoropyrimidine monotherapy / Panitumumab | 0
  7th line: Fluoropyrimidine + (Leucovorin or Folinic Acid) / Bevacizumab | 0

ADVERSE EVENTS:
Time Frame: Time from treatment initiation (for mCRC) up to 31 December 2020
Description: Since this is a retrospective study only relevant adverse events (AEs) have been collected.
  Definition of relevant AE: AE leading to first-line treatment switch, dose adaptation or discontinuation, or leading to death.
  Relevant AEs were assessed by System Organ Class (SOC).
Arm/Group | Non Interventional
All-Cause Mortality (participants affected / at risk) | 206/255
Serious Adverse Events (participants affected / at risk) | 40/255
Other Adverse Events (participants affected / at risk) | 104/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Interventional (N=255)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7 (9)
Cardiac disorders (Cardiac disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 18 (26)
General disorders and administration site conditions (General disorders) | 4 (4)
Hepatobiliary disorders (Hepatobiliary disorders) | 3 (3)
Immune system disorders (Immune system disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 3 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Investigations (Investigations) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5)
Nervous system disorders (Nervous system disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vascular disorders (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Interventional (N=255)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 23 (24)
Cardiac disorders (Cardiac disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 37 (51)
General disorders and administration site conditions (General disorders) | 25 (28)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2)
Immune system disorders (Immune system disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Investigations (Investigations) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders (Nervous system disorders) | 42 (44)
Renal and urinary disorder (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 13 (15)
Vascular disorders (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04317599/Prot_SAP_000.pdf